CLINICAL TRIAL: NCT04223843
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center, Parallel Group Study to Compare the Efficacy of Inhaled Tiotropium + Olodaterol, Fixed Dose Combination (5 mcg/5mcg) vs. Placebo Delivered by Respimat Inhaler in Patients With Moderate to Severe COPD, Stratified by Peak Inspiratory Flow Rate [TRONARTO].
Brief Title: A Study to Test the Combination of Tiotropium and Olodaterol Using the Respimat® Inhaler in People With Chronic Obstructive Pulmonary Disease (COPD) Who Have Different Abilities to Inhale
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1237-0095; 2019-001719-21 (EudraCT Number)
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Results first posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tiotropium-olodaterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Arm (Experimental): Tiotropium + Olodaterol Fixed Dose Combination (FDC) via Respimat
  Interventions: Drug: Tiotropium + olodaterol
- Placebo Arm (Placebo Comparator): Matching placebo via Respimat
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tiotropium + olodaterol — Oral Inhalation
  Arms: Active Arm
Drug: Placebo — Oral Inhalation
  Arms: Placebo Arm

SUMMARY:
To demonstrate the efficacy of inhaled tiotropium + olodaterol via Respimat® on lung function in patients with moderate to severe Chronic Obstructive Pulmonary Disease (COPD) with optimal and sub-optimal Peak Inspiratory Flow Rate (PIFR). Disease severity (moderate to severe) is based on the Global Initiative for Chronic Lung Disease (GOLD) guidelines (GOLD 2 - 3)

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent in accordance with International Council on Harmonisation Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
* Male or female patients, 40 years of age or older.
* All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria: patients with a post-bronchodilator Forced Expiratory Volume in one second (FEV1) >30% and <80% of predicted normal (European Coal and Steel Community (ECSC), [R94-1408]); and a postbronchodilator FEV1/ Functional Residual Capacity (FVC) <70%, at the screening visit.
* Patients must be current or ex-smokers with a smoking history of more than 10 pack years
* Patients should meet the peak inspiratory flow rate criteria (optimal or sub-optimal) at the time of randomization depending on which strata is available for inclusion in the study.
* Women of childbearing potential must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.
* Patients are expected to be able to perform, according to investigator's judgment, all trial related procedures including:

  * Technically acceptable pulmonary function tests (spirometry)
  * Use of In-Check DIAL G16 device to measure peak inspiratory flow rate.
  * Inhale medication in a competent manner (in the opinion of the investigator) from the Respimat® device
  * Perform technically acceptable body plethysmography measurements. This is applicable only to patients who will consent to the optional trial procedure at the selected sites.

Exclusion Criteria:

* Patients with a significant disease other than chronic obstructive pulmonary disease; a significant disease defined as a disease which, in the opinion of the investigator, and referring to the warnings to be observed as quoted in the locally applicable SmPC or prescribing information, could (i) put the patient at risk because of participation in the trial, (ii) influence the results of the trial, or (iii) cause concern regarding the patient's ability to participate in the trial.
* Patients who have had a chronic obstructive pulmonary disease exacerbation that required treatment with antibiotics, systemic steroids (oral or intravenous) or hospitalization in the 6 weeks prior to screening visit or during the screening period.
* Patients who experienced two or more moderate chronic obstructive pulmonary disease exacerbations (exacerbation that required treatment with antibiotics and/or oral corticosteroids), or one or more exacerbation leading to hospitalization within a year prior to visit 1.
* Patients with a history of asthma. For patients with allergic rhinitis or atopy, source documentation is required to verify that the patient does not have asthma.
* Patients taking inhaled corticosteroids (including combinations, e.g. inhaled corticosteroids / Long-Acting β2-agonist) in the 6 months prior to screening visit.
* Patients being treated with oral corticosteroid medication due to reasons other than chronic obstructive pulmonary disease exacerbation within 6 weeks prior to the screening visit.
* Patients who have completed a pulmonary rehabilitation program in the 6 weeks prior to screening visit or patients who are currently in a pulmonary rehabilitation program.
* Further criteria apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (21):
  - SEC Lung, Andalusia, Alabama
  - Jasper Summit Research, LLC, Jasper, Alabama
  - Meris Clinical Research, Brandon, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Clinical Research Specialists LLC, Kissimmee, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Best Clinical Trials, LLC, New Orleans, Louisiana
  - Infinity Medical Research, North Dartmouth, Massachusetts
  - Pulmonary Rsrch Inst of SE MI, Farmington Hills, Michigan
  - Minnesota Lung Center and Sleep Institute, Edina, Minnesota
  - Minnesota Lung Center, Woodbury, Minnesota
  - Valley Regional Hospital, Claremont, New Hampshire
  - CHEAR Center LLC, The Bronx, New York
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - Bernstein Clinical Rsrch Ctr, Cincinnati, Ohio
  - Lowcountry Lung and Critical Care, Charleston, South Carolina
  - Carolina Medical Research, Clinton, South Carolina
  - VitaLink Research -Gaffney, Gaffney, South Carolina
  - Vitalink Research - Spartansburg, Spartanburg, South Carolina
  - Diagnostics Research Group, San Antonio, Texas
- Germany (5):
  - Klinische Forschung Berlin GbR, Berlin
  - IKF Pneumologie GmbH & Co. KG, Frankfurt
  - Pneumologisches Forschungsinstitut an der LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Hamburger Institut für Therapieforschung GmbH (HIT), Hamburg
  - KLB Gesundheitsforschung Lübeck GmbH, Lübeck

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website. The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomised, double-blind, placebo-controlled trial to demonstrate the efficacy of 5µg/5µg inhaled tiotropium + olodaterol (Tio+Olo) via Respimat® on lung function in patients with moderate to severe chronic obstructive pulmonary disease (COPD) with optimal and sub-optimal peak inspiratory flow rate (PIFR).
Pre-assignment Details: Only patients that met all inclusion and none of the exclusion criteria were included in this trial. Prior to the initiation of any trial-related procedure, all patients were informed about the trial verbally and in writing by the investigator. Each patient signed and dated an Informed Consent Form (ICF) according to the local regulatory and legal requirements.
Groups:
- Tio+Olo (5μg/5μg) - Sub-optimal PIFR: A fixed dose combination of 5 microgram (μg)/5μg (two times 2.5µg/2.5µg) tiotropium + olodaterol (Tio+Olo) inhalation solution was administered orally once daily via Respimat inhaler in patients with moderate to severe chronic obstructive pulmonary disease (COPD) and with sub-optimal peak inspiratory flow rate (PIFR) (<60 Liter(L)/minute (min)) over a 4-week treatment period.
- Matching Placebo - Sub-optimal PIFR: 2 inhalation solutions of matching placebo were administered orally once daily via Respimat inhaler in patients with moderate to severe chronic obstructive pulmonary disease (COPD) and with sub-optimal peak inspiratory flow rate (PIFR) (<60 L/min) over a 4-week treatment period.
- Tio+Olo (5μg/5μg ) - Optimal PIFR: A fixed dose combination of 5μg/5μg (two times 2.5µg/2.5µg) tiotropium + olodaterol (Tio+Olo) inhalation solution was administered orally once daily via Respimat inhaler in patients with moderate to severe chronic obstructive pulmonary disease (COPD) and with sub-optimal peak inspiratory flow rate (PIFR) (≥60 L/min) over a 4-week treatment period.
- Matching Placebo - Optimal PIFR: 2 inhalation solutions of matching placebo were administered orally once daily via Respimat inhaler in patients with moderate to severe chronic obstructive pulmonary disease (COPD) and with optimal peak inspiratory flow rate (PIFR) (≥60 L/min) over a 4-week treatment period.
Period: Overall Study
Arm/Group | Tio+Olo (5μg/5μg) - Sub-optimal PIFR | Matching Placebo - Sub-optimal PIFR | Tio+Olo (5μg/5μg ) - Optimal PIFR | Matching Placebo - Optimal PIFR
Started | 55 | 55 | 51 | 52
Completed | 55 | 55 | 51 | 52
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This patient set included all randomised patients who were dispensed trial medication and were documented to have taken any dose of trial medication. The TS was used for demographics and baseline disease characteristics, concomitant therapies, treatment exposure, and safety analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tio+Olo (5μg/5μg) - Sub-optimal PIFR | Matching Placebo - Sub-optimal PIFR | Tio+Olo (5μg/5μg ) - Optimal PIFR | Matching Placebo - Optimal PIFR | Total
Number analyzed (Participants) | 55 | 55 | 51 | 52 | 213
Age, Continuous [Mean (Standard Deviation); unit: Years] — Treated Set.
  Years | 64 (9.79) | 67.05 (7.54) | 62.80 (7.48) | 65.88 (7.43) | 64.96 (8.25)
Sex: Female, Male [Count of Participants; unit: Participants] — Treated Set.
  Participants
    Female | 28 | 37 | 24 | 20 | 109
    Male | 27 | 18 | 27 | 32 | 104
Race (NIH/OMB) [Count of Participants; unit: Participants] — Treated Set.
  Participants
    American Indian or Alaska Native | 2 | 1 | 0 | 0 | 3
    Asian | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 2 | 3 | 1 | 0 | 6
    White | 51 | 51 | 50 | 51 | 203
    More than one race | 0 | 0 | 0 | 1 | 1
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Forced Expiratory Volume in one second (FEV1) area under the curve from 0 to 3 hours (AUC0-3h) [Mean (Standard Deviation); unit: Liter (L)] — FEV1 AUC0-3 at baseline. The baseline value will be the measurement made prior to the first dosing at Visit 2. If there are more than one measurement of FEV1 available prior to randomization, the mean of the two pre-dose pulmonary function test measurements at Visit 2, prior to the administration of the first dose of the randomized treatment, is used as the baseline FEV1. The area under the curve (AUC) is calculated as the area under the curve from 0 to 3 hours at baseline using the trapezoidal rule, divided by 3 hours to report in liters. Population: Full Analysis Set (FAS): This patient set was nested within the TS and included all patients who had a baseline and at least 1 post-baseline measurement for at least 1 efficacy endpoint. Only patients with availble data for this endpoint were included.
  Liter (L)
    number analyzed (Participants) | 43 | 47 | 44 | 47 | 181
    (all) | 1.224 (0.060) | 1.277 (0.079) | 1.388 (0.070) | 1.523 (0.074) | 1.324 (0.467)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1) Area Under the Curve From 0 to 3 Hours (AUC0-3h) After 4 Weeks of Treatment.
Description: FEV1 AUC0-3h was calculated as the area under the FEV1-time curve from 0 to 3h post-dose using the trapezoidal rule, divided by the duration (3h) to report in liters. Mean is adjusted mean.
  A hierarchical testing procedure was used to test the primary endpoint. Each of the tests were considered confirmatory only if all previous tests were successful.
Time Frame: At baseline and at week 4: 10 minutes (min) prior and 5 min, 15 min, 30 min and 1 hour (h), 2h and 3h after drug administration, respectively.
Population: Full Analysis Set (FAS): This patient set was nested within the TS and included all patients who had a baseline and at least 1 post-baseline measurement for at least 1 efficacy endpoint. Only patients with non-missing endpoint results were included.
Measure: Mean (Standard Error); unit: Liter (L)
Arm/Group | Tio+Olo (5μg/5μg) - Sub-optimal PIFR | Matching Placebo - Sub-optimal PIFR | Tio+Olo (5μg/5μg ) - Optimal PIFR | Matching Placebo - Optimal PIFR
Number analyzed (Participants) | 43 | 47 | 44 | 47
Liter (L) | 0.250 (0.033) | -0.086 (0.031) | 0.333 (0.032) | 0.012 (0.031)
Statistical Analysis 1: Comparison: Tio+Olo (5μg/5μg) - Sub-optimal PIFR vs Matching Placebo - Sub-optimal PIFR; H0: There is no difference in the mean FEV1 AUC0-3 change from baseline between Tio+Olo and matching placebo; Test type: Other; p < 0.0001, ANCOVA; Model included fixed categorical effects of treatment and the fixed continous effect of baseline FEV1 AUC0-3; Difference of adjusted means = 0.336, 95% CI 2-sided [0.246 to 0.425], Standard Error of Mean 0.045 — Difference = (Tio+Olo) - (Placebo)
Statistical Analysis 2: Comparison: Tio+Olo (5μg/5μg ) - Optimal PIFR vs Matching Placebo - Optimal PIFR; H0: There is no difference in the mean FEV1 AUC0-3h change from baseline between Tio+Olo and matching placebo; Test type: Other; p < 0.0001, ANCOVA; Model included the fixed categorical effect of treatment and the fixed continuous effect of baseline FEV1 AUC0-3h; Difference of adjusted means = 0.321, 95% CI 2-sided [0.233 to 0.409], Standard Error of Mean 0.044 — Difference = (Tio+Olo) - (Placebo)

2. Secondary Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1) After 4 Weeks of Treatment
Description: Change from baseline in trough Forced Expiratory Volume in one second (FEV1) after 4 weeks of treatment.
Time Frame: At baseline and at week 4.
Population: FAS: This patient set was nested within the TS and included all patients who had a baseline and at least 1 post-baseline measurement for at least 1 efficacy endpoint. Only patients with non-missing endpoint results were included.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Tio+Olo (5μg/5μg) - Sub-optimal PIFR | Matching Placebo - Sub-optimal PIFR | Tio+Olo (5μg/5μg ) - Optimal PIFR | Matching Placebo - Optimal PIFR
Number analyzed (Participants) | 50 | 52 | 47 | 50
Liter | 0.095 (0.031) | -0.106 (0.030) | 0.177 (0.030) | -0.040 (0.029)
Statistical Analysis 1: Comparison: Tio+Olo (5μg/5μg) - Sub-optimal PIFR vs Matching Placebo - Sub-optimal PIFR; H0: There is no difference in the mean trough FEV1 change from baseline between Tio+Olo and matching placebo; Test type: Other; p < 0.0001, Mixed Models Analysis; Mixed model with repeated measures including fixed categorial effect of treatment at each visit and fixed continuous effect of baseline at each visit; Difference of adjusted means = 0.201, 95% CI 2-sided [0.117 to 0.286], Standard Error of Mean 0.043 — Difference = (Tio+Olo) - (Placebo)
Statistical Analysis 2: Comparison: Tio+Olo (5μg/5μg ) - Optimal PIFR vs Matching Placebo - Optimal PIFR; H0: There is no difference in the mean trough FEV1 change from baseline between Tio+Olo and matching placebo; Test type: Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Difference of adjusted means = 0.217, 95% CI 2-sided [0.135 to 0.299], Standard Error of Mean 0.041 — Difference = (Tio+Olo) - (Placebo)

ADVERSE EVENTS:
Time Frame: From first intake of trial medication until last trial medication intake plus 21 days (residual effect period), up to 50 days.
Description: Treated Set: This patient set included all randomised patients who were dispensed trial medication and were documented to have taken any dose of trial medication. Adverse events were summarized by treatment group (Tio/Olo vs. Placebo), as defined in the statistical analysis plan.
Groups:
- 5μg/5μg Tio+Olo - Overall: A fixed dose combination (FDC) of 5μg/5μg (two times 2.5µg/2.5µg) tiotropium + olodaterol (Tio+Olo) inhalation solution was administered orally once daily via Respimat inhaler in patients with moderate to severe chronic obstructive pulmonary disease (COPD) over a 4-week treatment period. Overall group included patients with both, sub-optimal (<60 L/min) peak inspiratory flow rate (PIFR) and optimal (≥60 L/min) peak inspiratory flow rate (PIFR).
- Matching Placebo - Overall: 2 inhalation solutions of matching placebo were administered orally once daily via Respimat inhaler in patients with moderate to severe chronic obstructive pulmonary disease (COPD) over a 4-week treatment period. Overall group included patients with both, sub-optimal (<60 L/min) peak inspiratory flow rate (PIFR) and optimal (≥60 L/min) peak inspiratory flow rate (PIFR).
Arm/Group | 5μg/5μg Tio+Olo - Overall | Matching Placebo - Overall
All-Cause Mortality (participants affected / at risk) | 0/106 | 0/107
Serious Adverse Events (participants affected / at risk) | 2/106 | 1/107
Other Adverse Events (participants affected / at risk) | 0/106 | 0/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5μg/5μg Tio+Olo - Overall (N=106) | Matching Placebo - Overall (N=107)
Gastroenteritis (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/43/NCT04223843/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/43/NCT04223843/SAP_001.pdf